CLINICAL TRIAL: NCT01894321
Title: The Percutaneous Cholecystostomy is Appropriate as the Ultimate Treatment of Acute Cholecystitis in Critically Ill Patients: a Cross-sectional Study at Single Center.
Brief Title: The Clinical Outcomes of the Percutaneous Cholecystostomy, Supportive Care Versus Cholecystectomy.
Status: Completed | Type: Observational
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Byung Hyo Cha, MD, Medical Doctor, Cheju Halla General Hospital
Other Study IDs: PTGBD1
Record Dates: First submitted 2013-06-29; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Acute Calculous Cholecystitis; Acute Acalculous Cholecystitis
Keywords: Acute cholecystitis; Elderly; Critically ill patients; Surgical high risk; Percutaneous cholecystostomy; Cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous cholecystostomy (PC) is an effective treatment for cholecystitis in surgical high risk patients. However, there has been no definite agreement of the additional cholecystectomy in these patients. The investigators surveyed the clinical outcomes of the PC in surgical high risk patients. And the investigators tried to prove the PC can be appropriate and ultimate treatment for acute cholecystitis patients with critical illness through this study.

DETAILED DESCRIPTION:
Between 2007 and 2012, all patients admitted for acute cholecystitis, and then underwent ultrasonography guided percutaneous cholecystostomy in Cheju Halla General Hospital were consecutively enrolled.

Among 82 patients, 35 were performed laparoscopic cholecystectomy after recovery (Cholecystectomy group) and 47 treated by best supportive care without additional surgery (BSC group).

The investigators analyzed their surgical risks and clinical outcomes of both patients retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute cholecystitis
* Underwent the ultrasound-guided percutaneous cholecystostomy

Exclusion Criteria:

* Transferred patients from other institute after cholecystostomy procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From November 2007 to November 2012, patients admitted with acute cholecystitis through emergency center or out-patient clinic then underwent ultrasonography guided percutaneous cholecystostomy in Cheju Halla General Hospital were enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | within 30 days

SECONDARY OUTCOMES:
Evidence of recurrent cholecystitis or biliary complication | Within 30 days
  Acute cholecysitits : fever, abdominal pain, abnormal chemistry results Biliary complication : Gallstone pancreatitis, gallstone ileus or cholangitis
Evidence of recurrent cholecystitis or biliary complication | Within 30 days
  Acute cholecystits : fever, abdominal pain, abnormal chemistry results Biliary complication : Gallstone pancreatitis, gallstone ileus or cholangitis

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive disease center, Department of Internal Medicine, Cheju Halla General Hospital, Jeju City, Jeju Special Self-governing Province, South Korea

REFERENCES:
- [Background] Everhart JE, Khare M, Hill M, Maurer KR. Prevalence and ethnic differences in gallbladder disease in the United States. Gastroenterology. 1999 Sep;117(3):632-9. doi: 10.1016/s0016-5085(99)70456-7. PMID 10464139
- [Background] Kalliafas S, Ziegler DW, Flancbaum L, Choban PS. Acute acalculous cholecystitis: incidence, risk factors, diagnosis, and outcome. Am Surg. 1998 May;64(5):471-5. PMID 9585788
- [Background] Kiviluoto T, Siren J, Luukkonen P, Kivilaakso E. Randomised trial of laparoscopic versus open cholecystectomy for acute and gangrenous cholecystitis. Lancet. 1998 Jan 31;351(9099):321-5. doi: 10.1016/S0140-6736(97)08447-X. PMID 9652612
- [Background] Lo CM, Liu CL, Fan ST, Lai EC, Wong J. Prospective randomized study of early versus delayed laparoscopic cholecystectomy for acute cholecystitis. Ann Surg. 1998 Apr;227(4):461-7. doi: 10.1097/00000658-199804000-00001. PMID 9563529
- [Background] Koo KP, Thirlby RC. Laparoscopic cholecystectomy in acute cholecystitis. What is the optimal timing for operation? Arch Surg. 1996 May;131(5):540-4; discussion 544-5. doi: 10.1001/archsurg.1996.01430170086016. PMID 8624202
- [Background] Lujan JA, Parrilla P, Robles R, Marin P, Torralba JA, Garcia-Ayllon J. Laparoscopic cholecystectomy vs open cholecystectomy in the treatment of acute cholecystitis: a prospective study. Arch Surg. 1998 Feb;133(2):173-5. doi: 10.1001/archsurg.133.2.173. PMID 9484730
- [Background] Houghton PW, Jenkinson LR, Donaldson LA. Cholecystectomy in the elderly: a prospective study. Br J Surg. 1985 Mar;72(3):220-2. doi: 10.1002/bjs.1800720327. PMID 3978383
- [Background] Frazee RC, Nagorney DM, Mucha P Jr. Acute acalculous cholecystitis. Mayo Clin Proc. 1989 Feb;64(2):163-7. doi: 10.1016/s0025-6196(12)65670-5. PMID 2921875
- [Background] Weiss CA 3rd, Lakshman TV, Schwartz RW. Current diagnosis and treatment of cholecystitis. Curr Surg. 2002 Jan-Feb;59(1):51-4. doi: 10.1016/s0149-7944(01)00628-6. No abstract available. PMID 16093104
- [Background] Vogelzang RL, Nemcek AA Jr. Percutaneous cholecystostomy: diagnostic and therapeutic efficacy. Radiology. 1988 Jul;168(1):29-34. doi: 10.1148/radiology.168.1.3289094.
- [Background] Hultman CS, Herbst CA, McCall JM, Mauro MA. The efficacy of percutaneous cholecystostomy in critically ill patients. Am Surg. 1996 Apr;62(4):263-9. PMID 8600844
- [Background] Welschbillig-Meunier K, Pessaux P, Lebigot J, Lermite E, Aube Ch, Brehant O, Hamy A, Arnaud JP. Percutaneous cholecystostomy for high-risk patients with acute cholecystitis. Surg Endosc. 2005 Sep;19(9):1256-9. doi: 10.1007/s00464-004-2248-6. Epub 2005 Jul 14. PMID 16132331
- [Background] Byrne MF, Suhocki P, Mitchell RM, Pappas TN, Stiffler HL, Jowell PS, Branch MS, Baillie J. Percutaneous cholecystostomy in patients with acute cholecystitis: experience of 45 patients at a US referral center. J Am Coll Surg. 2003 Aug;197(2):206-11. doi: 10.1016/S1072-7515(03)00143-1. PMID 12892798
- [Background] Hirota M, Takada T, Kawarada Y, Nimura Y, Miura F, Hirata K, Mayumi T, Yoshida M, Strasberg S, Pitt H, Gadacz TR, de Santibanes E, Gouma DJ, Solomkin JS, Belghiti J, Neuhaus H, Buchler MW, Fan ST, Ker CG, Padbury RT, Liau KH, Hilvano SC, Belli G, Windsor JA, Dervenis C. Diagnostic criteria and severity assessment of acute cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):78-82. doi: 10.1007/s00534-006-1159-4. Epub 2007 Jan 30. PMID 17252300
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Hatzidakis AA, Prassopoulos P, Petinarakis I, Sanidas E, Chrysos E, Chalkiadakis G, Tsiftsis D, Gourtsoyiannis NC. Acute cholecystitis in high-risk patients: percutaneous cholecystostomy vs conservative treatment. Eur Radiol. 2002 Jul;12(7):1778-84. doi: 10.1007/s00330-001-1247-4. Epub 2002 Feb 21. PMID 12111069
- [Background] Escarce JJ, Shea JA, Chen W, Qian Z, Schwartz JS. Outcomes of open cholecystectomy in the elderly: a longitudinal analysis of 21,000 cases in the prelaparoscopic era. Surgery. 1995 Feb;117(2):156-64. doi: 10.1016/s0039-6060(05)80079-0. PMID 7846619
- [Background] Morse BC, Smith JB, Lawdahl RB, Roettger RH. Management of acute cholecystitis in critically ill patients: contemporary role for cholecystostomy and subsequent cholecystectomy. Am Surg. 2010 Jul;76(7):708-12. doi: 10.1177/000313481007600724. PMID 20698375
- [Background] McKay A, Abulfaraj M, Lipschitz J. Short- and long-term outcomes following percutaneous cholecystostomy for acute cholecystitis in high-risk patients. Surg Endosc. 2012 May;26(5):1343-51. doi: 10.1007/s00464-011-2035-0. Epub 2011 Nov 17. PMID 22089258
- [Background] Granlund A, Karlson BM, Elvin A, Rasmussen I. Ultrasound-guided percutaneous cholecystostomy in high-risk surgical patients. Langenbecks Arch Surg. 2001 Apr;386(3):212-7. doi: 10.1007/s004230100211. PMID 11382324
- [Background] Ha JP, Tsui KK, Tang CN, Siu WT, Fung KH, Li MK. Cholecystectomy or not after percutaneous cholecystostomy for acute calculous cholecystitis in high-risk patients. Hepatogastroenterology. 2008 Sep-Oct;55(86-87):1497-502. PMID 19102330
- [Background] Leveau P, Andersson E, Carlgren I, Willner J, Andersson R. Percutaneous cholecystostomy: a bridge to surgery or definite management of acute cholecystitis in high-risk patients? Scand J Gastroenterol. 2008;43(5):593-6. doi: 10.1080/00365520701851673. PMID 18415753
- [Background] Bakkaloglu H, Yanar H, Guloglu R, Taviloglu K, Tunca F, Aksoy M, Ertekin C, Poyanli A. Ultrasound guided percutaneous cholecystostomy in high-risk patients for surgical intervention. World J Gastroenterol. 2006 Nov 28;12(44):7179-82. doi: 10.3748/wjg.v12.i44.7179. PMID 17131483
- [Background] Koebrugge B, van Leuken M, Ernst MF, van Munster I, Bosscha K. Percutaneous cholecystostomy in critically ill patients with a cholecystitis: a safe option. Dig Surg. 2010;27(5):417-21. doi: 10.1159/000308460. Epub 2010 Oct 15. PMID 20948216
- [Background] Chok KS, Chu FS, Cheung TT, Lam VW, Yuen WK, Ng KK, Chan SC, Poon RT, Yeung C, Lo CM, Fan ST. Results of percutaneous transhepatic cholecystostomy for high surgical risk patients with acute cholecystitis. ANZ J Surg. 2010 Apr;80(4):280-3. doi: 10.1111/j.1445-2197.2009.05105.x. PMID 20575957
- [Background] Griniatsos J, Petrou A, Pappas P, Revenas K, Karavokyros I, Michail OP, Tsigris C, Giannopoulos A, Felekouras E. Percutaneous cholecystostomy without interval cholecystectomy as definitive treatment of acute cholecystitis in elderly and critically ill patients. South Med J. 2008 Jun;101(6):586-90. doi: 10.1097/SMJ.0b013e3181757b77. PMID 18475218